CLINICAL TRIAL: NCT00806039
Title: Impact of EArly Renal Involvement on the Developement of Severe In-hospital Renal Failure
Brief Title: Impact of Early Renal Involvement on the Development of Severe In-hospital Renal Failure
Acronym: EARLI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint Louis VA Medical Center (U.S. Federal Agency)
Responsible Party: Tarek El-Achkar, MD, Saint Louis VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1143004
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Kidney Failure, Acute; Renal Insufficiency, Acute; Kidney Failure; Renal Insufficiency
Keywords: Kidney Failure, Acute; Renal Insufficiency, Acute; Kidney Failure; Renal Insufficiency
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Early renal involvement
  Interventions: Other: Early Renal Involvement
- 2 (No Intervention): control

INTERVENTIONS:
Other: Early Renal Involvement — Renal Consultation
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether renal team involvement early at the onset of kidney injury will prevent further developement of more severe renal failure and worse hospitalization outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized, elevation in creatinine meeting definition

Exclusion Criteria:

* CDK5, ESRD,solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Severe renal Failure | 10 days

SECONDARY OUTCOMES:
Composite outcome morbidity mortality | hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M El-Achkar, MD, Study Director — Saint Louis VA Medical Center
Locations (1):
- Saint Louis VA Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Derived] Balasubramanian G, Al-Aly Z, Moiz A, Rauchman M, Zhang Z, Gopalakrishnan R, Balasubramanian S, El-Achkar TM. Early nephrologist involvement in hospital-acquired acute kidney injury: a pilot study. Am J Kidney Dis. 2011 Feb;57(2):228-34. doi: 10.1053/j.ajkd.2010.08.026. Epub 2010 Dec 31. PMID 21195518